CLINICAL TRIAL: NCT01696981
Title: Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial
Brief Title: Screening for Colorectal Cancer in Older Patients (PLCO Screening Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NCI-2012-01757; NCI-2012-01757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000078532; NCI-P93-0050; PLCO-1; PLCO-Colorectal (Other: National Cancer Institute)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Colon Carcinoma; Rectal Carcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Sigmoidoscopy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Colorectal Screening (Active Comparator): Participants undergo a colorectal examination with a flexible sigmoidoscope at baseline and year 5. Participants complete a DQX at baseline and DHQ at year 3. An ADU (previously referred to as the PSH questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident colorectal cancers as all deaths that occur among both screened and control subjects during the trial.
  Interventions: Other: Screening Questionnaire Administration; Procedure: Sigmoidoscopy
- Control (No Intervention): Participants receive standard medical care. Participants complete a DHQ at baseline.

INTERVENTIONS:
Other: Screening Questionnaire Administration — Undergo questionnaire assessments
  Arms: Colorectal Screening
Procedure: Sigmoidoscopy — Undergo a flexible sigmoidoscopy
  Other Names: Proctosigmoidoscopy
  Arms: Colorectal Screening

SUMMARY:
This clinical trial studies whether screening methods used to diagnose cancer of the prostate, lung, colon, rectum, or ovaries can reduce deaths from these cancers. Screening tests may help doctors find cancer cells early and plan better treatment for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether screening with flexible sigmoidoscopy (60-cm sigmoidoscope) can reduce mortality from colorectal cancer in women and men aged 55-74 at study entry.

SECONDARY OBJECTIVES:

I. To assess screening variables, other than mortality, for each of the interventions including sensitivity, specificity, and positive predictive value.

II. To assess the incidence, stage, and survival of cancer cases. III. To investigate the mortality predictive value of biologic and/or prognostic characterizations of tumor tissue as intermediate endpoints.

IV. To conduct biomolecular and genetic research into factors associated with cancer carcinogenesis and promotion, as well as the early detection of these factors.

OUTLINE: Participants in the overall PLCO study are stratified by screening center, gender, and age (55-59 vs 60-64 vs 65-69 vs 70-74). Participants are randomized to 1 of 2 arms (control vs screening).

ARM I (Control): Participants receive standard medical care. Participants complete a Diet History Questionnaire (DHQ) at baseline.

ARM II (Colorectal Screening): Participants undergo a colorectal examination with a flexible sigmoidoscope at baseline and year 5. A scheduling and tracking procedure is implemented to ensure regular attendance at repeat screens for participants screened negative or for those who are designated suspicious or positive at screening but for whom subsequent diagnostic procedures do not reveal colorectal cancer (follow-up diagnostic procedures are through their own medical care environment). Participants diagnosed with colorectal cancer via a screening test are referred for treatment in accordance with current accepted practice for appropriate stage of disease, patient age, and medical condition; a procedure is provided for contact with qualified medical personnel to insure appropriate therapy.

Participants complete a Dietary Questionnaire (DQX) at baseline and DHQ at year 3. An Annual Study Update (ADU) (previously referred to as the Periodic Survey of Health [PSH] questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident colorectal cancers as all deaths that occur among both screened and control subjects during the trial.

After completion of screening, participants are followed up for at least 13 years.

ELIGIBILITY:
Exclusion Criteria:

* Men and women who at the time of randomization are less than 55 or greater than or equal to 75 years of age
* Individuals undergoing treatment for cancer at this time, excluding basal-cell and squamous-cell skin cancer
* Individuals with known prior cancer of the colon, rectum, lung, prostate

  * This includes primary or metastatic PLCO cancers
* Individuals with previous surgical removal of the entire colon, one lung, or the entire prostate (men only)

  * Until October 1996, women with previous surgical removal of both ovaries were excluded from the trial. In order to increase the enrollment of women into the trial, beginning in October 1996, these women were no longer excluded for this reason.
* Individuals who are participating in another cancer screening or cancer primary prevention trial
* Males who have taken Proscar/Propecia/finasteride in the past 6 months

  * NOTE: Individuals who are already enrolled in the trial when their physician prescribes finasteride are not prevented from taking this medication. As a result, these participants will continue to be screened and followed just as those participants who are not on finasteride.
  * NOTE: Men who are taking Tamoxifen are not excluded from any part of the PLCO Screening Trial.
  * Prior to April 1, 1999 women were excluded from the trial if they were currently taking or had taken Tamoxifen or Evista\Raloxifene in the past 6 months. As of April 1999 based on a decision from the PLCO Ovary Subcommittee, women who have or are currently taking Tamoxifen or Evista\Raloxifene are not excluded from participation.
* Individuals who are unwilling or unable to sign the informed consent form
* Males who have had more than one PSA blood test in the past three years
* Individuals who have had a colonoscopy, sigmoidoscopy, or barium enema in the past three years

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154900 (Actual)
Dates: Start 1993-11-16 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine D Berg, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Malcomson FC, Shams-White MM, Reedy J, Huang WY, Moore SC, Loftfield E. Adherence to the 2018 World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Recommendations and risk of lifestyle-related cancers in the prostate, lung, colorectal, and ovarian cancer screening trial. BJC Rep. 2025 Nov 19;3(1):81. doi: 10.1038/s44276-025-00195-6. PMID 41261199
- [Derived] Fan Z, Zhang Y, Yao Q, Liu X, Duan H, Liu Y, Sheng C, Lyu Z, Yang L, Song F, Huang Y, Song F. Effects of joint screening for prostate, lung, colorectal, and ovarian cancer - results from a controlled trial. Front Oncol. 2024 Apr 29;14:1322044. doi: 10.3389/fonc.2024.1322044. eCollection 2024. PMID 38741776
- [Derived] Jiang Y, Xie Q, Chen R. Breast Cancer Incidence and Mortality in Relation to Hormone Replacement Therapy Use Among Postmenopausal Women: Results From a Prospective Cohort Study. Clin Breast Cancer. 2022 Feb;22(2):e206-e213. doi: 10.1016/j.clbc.2021.06.010. Epub 2021 Jun 26. PMID 34548240
- [Derived] Wang K, Wu Q, Li Z, Reger MK, Xiong Y, Zhong G, Li Q, Zhang X, Li H, Foukakis T, Xiang T, Zhang J, Ren G. Vitamin K intake and breast cancer incidence and death: results from a prospective cohort study. Clin Nutr. 2021 May;40(5):3370-3378. doi: 10.1016/j.clnu.2020.11.009. Epub 2020 Nov 16. PMID 33277073
- [Derived] Kunzmann AT, Coleman HG, Huang WY, Cantwell MM, Kitahara CM, Berndt SI. Fruit and vegetable intakes and risk of colorectal cancer and incident and recurrent adenomas in the PLCO cancer screening trial. Int J Cancer. 2016 Apr 15;138(8):1851-61. doi: 10.1002/ijc.29922. Epub 2015 Dec 8. PMID 26559156
- [Derived] Kunzmann AT, Coleman HG, Huang WY, Kitahara CM, Cantwell MM, Berndt SI. Dietary fiber intake and risk of colorectal cancer and incident and recurrent adenoma in the Prostate, Lung, Colorectal, and Ovarian Cancer Screening Trial. Am J Clin Nutr. 2015 Oct;102(4):881-90. doi: 10.3945/ajcn.115.113282. Epub 2015 Aug 12. PMID 26269366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between November 1993 and July 2001 at 10 study centers. Recruitment was done for all four outcomes of the study (prostate, lung, colorectal and ovarian).
Pre-assignment Details: Participants signed a study informed consent prior to being randomized to a study arm.
Groups:
- Control: Participants receive standard medical care. Participants complete a baseline questionnaire at entry and a dietary history questionnaire (DHQ) during study years 0-6.
- Colorectal Screening: Participants undergo a colorectal examination with a flexible sigmoidoscope at baseline and year 5. Participants complete a Dietary Questionnaire (DQX) at baseline and a Dietary History Questionnaire (DHQ) at study years 3-6. An Annual Study Update (ASU) (previously referred to as the Periodic Survey of Health [PSH] questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident colorectal cancers and all deaths that occur among both screened and control arm subjects during the trial.
Period: Overall Study
Arm/Group | Control | Colorectal Screening
Started | 77455 | 77445
Completed | 76254 | 67071
Not Completed | 1201 | 10374
Not completed — Cancer Before Rand. (Colo. Screening) | 0 | 20
Not completed — Died Before Randomization | 3 | 8
Not completed — Died Before ASU (Control) | 278 | 0
Not completed — Refused ASU (Control) | 920 | 0
Not completed — Refused Screen (Colorectal Screening) | 0 | 10346

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Colorectal Screening | Total
Number analyzed (Participants) | 77455 | 77445 | 154900
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49610 | 49634 | 99244
  >=65 years | 27845 | 27811 | 55656
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (5.4) | 62.6 (5.4) | 62.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39111 | 39105 | 78216
  Male | 38344 | 38340 | 76684
Region of Enrollment [Number; unit: participants]
  United States | 77455 | 77445 | 154900

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Deaths
Description: Colorectal cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Measure: Number; unit: Participants
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Participants | 341 | 252

2. Secondary Outcome: Deaths From All Causes
Description: Deaths from all causes were compared between the colorectal cancer screening arm and the usual care arm.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Population: All participants. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Participants | 11064 | 10835

3. Secondary Outcome: Death Rates From All Causes
Description: Deaths from all causes were compared between the colorectal cancer screening arm and the usual care arm. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Population: All participants. An intention-to-treat analysis was performed.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Deaths per 10,000 PY | 127.0 | 124.3
Statistical Analysis 1: Comparison: Control vs Colorectal Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.95 to 1.00]

4. Secondary Outcome: Colorectal Cancer Incidence
Description: Colorectal cancer diagnoses confirmed by medical record abstraction.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Population: All participants. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Participants | 1287 | 1012

5. Secondary Outcome: Colorectal Cancer Incidence Rates
Description: Colorectal cancer diagnoses confirmed by medical record abstraction. Incidence rate (cumulative) defined as colorectal cancer diagnoses divided by person years at risk for colorectal cancer.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Population: All participants. An intention-to-treat analysis was performed.
Measure: Number; unit: Diagnoses per 10,000 PY
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Diagnoses per 10,000 PY | 15.2 | 11.9
Statistical Analysis 1: Comparison: Control vs Colorectal Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.72 to 0.85]

6. Secondary Outcome: Complications of Diagnostic Evaluation Following a Positive Screening Test
Description: Number of participants who experienced complications during diagnostic work-up of a positive colorectal examination.
Time Frame: One year from screening examination
Population: The units analyzed were positive screening exams with documented diagnostic follow-up. If a participant received 2 positive screens with documented follow-up after each one, he would be counted 2 times in the number of units analyzed.
Measure: Number; unit: Positive screens w/ complications
Units Other Than Participants: Positive Screens with Follow-up
Arm/Group | Colorectal Screening
Number analyzed (Participants) | 21896
Number analyzed (Positive Screens with Follow-up) | 24976
Positive screens w/ complications
  When DE Led to Colorectal Cancer Diagnosis | 58
  When DE Did Not Lead to Colorectal Cancer Diag | 279

7. Primary Outcome: Colorectal Cancer Death Rates
Description: Colorectal cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.1 years.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Colorectal Screening
Number analyzed (Participants) | 77455 | 77445
Deaths per 10,000 PY | 3.9 | 2.9
Statistical Analysis 1: Comparison: Control vs Colorectal Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.87]

8. Secondary Outcome: T0 (Baseline) FSG Screening Results
Description: Flexible sigmoidoscopy (FSG) result
Time Frame: T0 (at study entry)
Population: All participants in the Colorectal Screening arm who had an FSG at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Colorectal Screening
Number analyzed (Participants) | 64653
Participants
  Negative | 42403
  Positive | 15154
  Inadequate screen | 7096

9. Secondary Outcome: T3/T5 FSG Screening Result
Description: Flexible sigmoidoscopy (FSG) result
Time Frame: T3 (three years after entry) or T5 (five years after entry)
Population: All participants in the Colorectal Screening arm who had an FSG at T0 or T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Colorectal Screening
Number analyzed (Participants) | 41858
Participants
  Negative | 26694
  Positive | 9818
  Inadequate screen | 5346

ADVERSE EVENTS:
Time Frame: During each annual screening visit.
Description: These events are solely those prompted by the screening examination.
Arm/Group | Colorectal Screening
Serious Adverse Events (participants affected / at risk) | 0/77445
Other Adverse Events (participants affected / at risk) | 504/77445
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Screening (N=77445)
Anxiety (General disorders) | 2 (2)
Bleeding (General disorders) | 53 (53)
Dizzy (General disorders) | 204 (210)
Fainted (General disorders) | 101 (101)
Nausea (General disorders) | 101 (101)
Pain (General disorders) | 41 (42)
Perforated Bowel (General disorders) | 3 (3)
Other Adverse Event (General disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less